CLINICAL TRIAL: NCT06200740
Title: Remotely Observed Methadone Evaluation (ROME)
Brief Title: Remotely Observed Methadone Evaluation
Acronym: ROME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonara Health (Industry)
Collaborators: Oregon Health and Science University (Other); Stanford University (Other); Adapt Oregon (Unknown)
Responsible Party: Principal Investigator, Michael Giles, Chief Executive Officer, Sonara Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VDW001; R43DA056259 (NIH)
Record Dates: First submitted 2023-12-08; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Sonara — web application facilitating asynchronous observation of methadone dosing
  Other Names: Elpida; Virtual dosing window

SUMMARY:
Opioid addiction, which affects 16 million individuals worldwide, can be treated using methadone, a proven and effective opioid medication for treating OUD that extends retention in care, reduces mortality, and inhibits illicit drug use. However, methadone treatment is limited to federally certified Opioid Treatment Programs (OTPs), which must meet complex regulatory requirements, and require new patients to take their dose in person six days per week, presenting significant barriers to treatment. To address these barriers, Sonara Heath has developed the Sonara software platform, which will enable OTPs to offer accelerated take-home methadone regimens while maintaining safety and diversion prevention.

ELIGIBILITY:
Inclusion Criteria:

* Receiving methadone for the treatment of opioid use disorder

Exclusion Criteria:

* Patients with >13 take-homes
* Patients with positive toxicology results in last 30-60 days
* Patients involved with drug court ineligible for take-homes
* Patients without adequate access to technology
* Patients with <30 days in treatment
* Patients with mental health instability
* Patients with recent diversion attempts
* Patients using buprenorphine for agonist therapy
* Patients guest dosing at another clinic during trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | two weeks
  The SUS, a 10-item scale with each item rated on a 5-point scale (scored 0 to 4) with five negative statements (e.g., system is unnecessarily complex) (reverse scored) and five positive statements (e.g., system functions are well integrated), evaluated user perceptions of the system's usability. We summed scores and multiplied them by 2.5 for the total score with a range from 0 to 100 (Lewis, 2018).

SECONDARY OUTCOMES:
Acceptability, Appropriateness and Feasibility of Implementation Measures | two weeks
  Acceptability Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) are single factor 4-item scales scored 1 to 5 and summed with test-retest reliabilities of 0.73 to 0.88 (Weiner et al., 2017). Scores for each of the three dimensions have a potential range of 4 to 20 with higher scores suggesting better implementation potential.

CONTACTS AND LOCATIONS:
Locations (1):
- Adapt - Roseburg, Roseburg, Oregon, United States

IPD SHARING:
Plan to Share IPD: No